CLINICAL TRIAL: NCT06394804
Title: Combination Targeted and Hormonal treAtMEnt of Low-gradE Serous Ovarian Cancer in the upfroNt Setting
Brief Title: A Study of Avutometinib, Defactinib, and Letrozole in People With Low-Grade Serous Ovarian Cancer
Acronym: CHAMELEON
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-014
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Low-Grade Serous Ovarian Cancer
Keywords: Avutometinib; Defactinib; Letrozole; 24-014
MeSH Terms: interventions — defactinib; Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avutometinib, Defactinib, and Letrozole (Experimental): Enrolled patients will be treated with avutometinib 3.2 mg PO, twice weekly (e.g. M/Th,Tu/F, or W/Sa) + defactinib 200 mg PO BID for 3 weeks, followed by a 1 week rest period, in each 4-week (28 day) cycle. Patients will also be treated with letrozole 2.5 mg PO daily, and pre/perimenopausal patients will also receive leuprolide acetate 3.75 mg IM every 4 weeks or 11.25 mg every 3 months for ovarian suppression while an ovary remains in situ.
  Interventions: Drug: Avutometinib; Drug: Defactinib; Drug: Letrozole

INTERVENTIONS:
Drug: Avutometinib — Starting Dose 3.2 mg BIW for 3 of 4 weeks, Dose -1, 2.4 mg BIW for 3 of 4 weeks
  Other Names: VS-6766
Drug: Defactinib — Starting Dose 200 mg BID for 3 of 4 weeks, Dose -1, 200 mg QD for 3 of 4 weeks
  Other Names: VS-6063
Drug: Letrozole — 2.5 mg PO daily

SUMMARY:
The researchers are doing this study to find out whether the combination of avutometinib, defactinib, and letrozole is an effective treatment for people with low-grade serous ovarian cancer (LGSOC). The researchers will also look at the safety of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ≥ 18 years of age
* Histologically-confirmed LGSOC (ovarian, peritoneal) by tissue biopsy read by pathology at study institution. NOTE: Patients with a prior history of serous borderline tumors without prior systemic (cytotoxic or hormonal) treatment but a new diagnosis of low-grade serous ovarian cancer are eligible.
* Determination that the patient is not a primary surgical candidate by a gynecologic oncologist surgeon; or has undergone an attempted primary debulking with residual RECIST measurable disease.
* Measurable disease according to RECIST 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension. Each lesion must be ≥10mm when measured by CT or MRI. Lymph nodes must be ≥15mm by short axis when measured by CT or MRI.
* An Eastern Cooperative Group (ECOG) performance status of ≤1. Patients with an ECOG performance status of 2 are permitted on trial if this is deemed to be secondary to cancer but not to other comorbidities.
* Patients with treated brain metastases are eligible if follow-up brain imaging after CNS-directed therapy shows no evidence of progression. Patients with asymptomatic brain metastases that do not require intervention are also eligible.
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on anti-HCV treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Female patients with reproductive potential agree to use highly effective method of contraceptive during the trial and for 1 month following the last dose of study intervention, unless surgical menopause is conferred. Women of child-bearing potential must have a negative pregnancy test within 14 days prior to commencement of study treatment. Non-hormonal methods of highly effective contraception include:

  * intrauterine device (IUD)
  * bilateral tubal occlusion
  * vasectomized partner
  * sexual abstinence
* Patients must have adequate cardiac function with left ventricular ejection fraction ≥ 50% by echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan.
* Baseline QTc interval < 460 ms (Common Terminology Criteria for Adverse Events [CTCAE] Grade 1) using Fredericia's QT correction formula. NOTE: This criterion does not apply to patients with a right or left bundle branch block.
* Adequate organ function, defined by the following parameters:

  °Adequate hematologic function
* Hemoglobin [Hb] ≥ 9.0 g/dL. If a red blood cell transfusion has been administered the Hb must remain stable and ≥ 9.0 g/dL for at least 1 week prior to first dose of study intervention.
* Platelets ≥ 100,000/mm^3
* Absolute neutrophil count [ANC] ≥ 1000/mm^3

  °Adequate hepatic function:
* Total bilirubin ≤1.5 × upper limit of normal [ULN] for the institution; patients with Gilbert syndrome may enroll if total bilirubin is <3.0mg/dL (51 μmole/L) upon discussion with MSK PI.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (or <5 xULN in patients with liver metastases).

  * Adequate renal function with creatinine clearance rate of ≥50 mL/min as calculated by the Cockcroft-Gault formula or serum creatinine of ≤ 1.5 x ULN.
  * Creatine phosphokinase (CPK) ≤2.5 x ULN.

Exclusion Criteria:

* Patients who are deemed in the opinion of their treating physician to be appropriate candidates for a primary debulking surgery are not eligible for this trial, unless measurable disease remains after a primary cytoreductive surgery.
* Prior systemic anti-cancer therapy for LGSOC or serous borderline disease.
* Major surgery within 4 weeks, minor surgery within 2 weeks, or palliative radiotherapy within 1 week of the first dose of study intervention. Open and close laparotomy and/or laparoscopy will be considered minor surgery.
* Treatment with warfarin. Patients on warfarin for deep vein thrombosis/pulmonary embolism can be converted to low-molecular-weight heparin or direct oral anticoagulants (DOACs).
* Patients with the inability to swallow oral medications or impaired gastrointestinal absorption due to gastrectomy or drainage PEG tube. Patients with diagnosis of bowel obstruction <3 months from study enrollment will be excluded unless surgically cured or approved by study PI.
* Symptomatic brain metastases requiring steroids or other interventions. Patients with new asymptomatic CNS metastases detected during the screening period must receive radiation therapy and/or surgery for CNS metastases. Following treatment, these patients may then be eligible if all other criteria are met.
* Patients with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
* Patients with a history of corneal erosion (instability of corneal epithelium), corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions.
* History of rhabdomyolysis.
* Patients with a history of hypersensitivity to any of the active (Avutometinib, defactinib) or inactive (hydroxypropylmethylcellulose, mannitol, magnesium stearate) ingredients of the investigational product.
* Female patients who are breastfeeding.
* Any other medical condition (e.g., cardiac, gastrointestinal, pulmonary, psychiatric, neurological, genetic, etc.) that in the opinion of the Investigator would places the patient at unacceptably high risk for toxicity.
* Exposure to medications (with or without prescriptions), supplements, herbal remedies, or foods with potential for drug-drug interactions with study interventions within 14 days prior to the first dose of study intervention and during the course of therapy (Appendix 1), including:

  * strong CYP3A4 inhibitors or inducers, due to potential drug-drug interactions with both Avutometinib and defactinib.
  * strong CYP2C9 inhibitors or inducers, due to potential drug-drug interactions with defactinib.
  * P-glycoprotein (P-gp) inhibitors or inducers, due to potential drug-drug interactions with defactinib.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer
Enrollment: 20 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 2 years
  as defined by complete response or partial response assessed by RECIST v1.1. in patients receiving neoadjuvant treatment or treatment for measurable disease following suboptimal debulking.

SECONDARY OUTCOMES:
Occurrence of adverse events | 2 years
  as assessed by CTCAE (Common Terminology Criteria for Adverse Events) v.5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Grisham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk -Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm